CLINICAL TRIAL: NCT06624280
Title: Does Orthopedic Surgery Improve Gait Efficiency in Children With Cerebral Palsy? A Retrospective Study
Acronym: OrthoSurg01
Status: Completed | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Principal Investigator, Silvia Faccioli, Principal Investigator, Azienda USL Reggio Emilia - IRCCS
Other Study IDs: 134/2023/OSS/AUSLRE
Record Dates: First submitted 2024-09-20; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Cerebral Palsy (CP)
Keywords: Cerebral palsy; Orthopedics; Gait Analysis; Child; Adolescent; Physically Challenged; Rehabilitation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SEMLS group: The study population will include patients who attended the Children Rehabilitation Unit of Local Health Authority of Reggio Emilia from 2011 to 2021. The study will focus on patients diagnosed with cerebral palsy who underwent lower limb SEMLS (single-event multilevel surgery) and 3D Gait Analysis before and after surgery.
  Interventions: Procedure: single-event multilevel surgery

INTERVENTIONS:
Procedure: single-event multilevel surgery — surgical orthopedic approach where multiple deformities are corrected in one solution, often involving both lower limbs, to improve walking performance

SUMMARY:
Purpose: The aim of this retrospective observational study is to describe the demographic, clinical, and functional characteristics of children and adolescents with spastic cerebral palsy (CP) undergoing Single Event Multilevel Surgery (SEMLS) and changes in their gait efficiency following surgery.

Methods: Seventy-eight participants were included and a total of eighty-four SEMLS analyzed. All the participants were followed by the Children Rehabilitation Unit of the Local Health Authority of Reggio Emilia. Participants met the following requirements: age 4-20 years; hemiplegic or diplegic CP; Gross Motor Function Classification System level I, II or III; 3D gait analysis either before and after surgery. The following parameters were reported: maximum hip and knee extension in the gait cycle, to measure the gait efficiency; normalized maximum power produced by the ankle during push-off phase, to express the propulsive capacity; normalized speed and normalized stride length as global gait performance measure.

DETAILED DESCRIPTION:
Children with Cerebral Palsy (CP) often have gait difficulties due to poor motor control, spasticity, skeletal deformities, and muscle weakness. Their walking is usually slow, tiring, with reduced endurance, and a higher risk of falls. As a result, these children often have limited participation in daily activities and a lower quality of life. Among the most common treatments, functional orthopedic surgery is now considered the "standard of care" for these patients. Many studies have shown that surgery has a positive impact on walking ability.

In the traditional surgical approach, patients undergo multiple operations, each correcting a single issue. For example, fixing a shortened triceps muscle, to allow the foot to fully contact the ground, might be followed by lengthening the knee flexors to enable full knee extension and upright standing. This step-by-step process, where surgeries are often done annually, was called the "birthday syndrome". Some researchers have studied the effects of surgery on specific walking issues. For example, in 2022, Kruger K.R. et al. examined the long-term impact of correcting valgus-pronated feet. Dohin B. et al., in 2020, looked at how lengthening knee flexors and adductors improved in-toeing gait. Krupiński M. et al., in 2015, studied the effect of Achilles tendon lengthening in children with toe-walking (equinus gait). While these studies provided useful insights for clinicians, they often oversimplified the complexity of the underlying problems.

In CP, multiple areas of the body are usually involved in walking difficulties, as seen in crouch gait (walking with bent knees), which can have many causes that influence each other. This often requires surgery on multiple areas at once to improve the overall balance of the body. More recently, surgeons have adopted a technique where multiple deformities are corrected in a single surgery, often involving both lower limbs. This approach, known as single-event multilevel surgery (SEMLS), reduces the number of surgeries compared to the traditional method of addressing one issue at a time. However, as children grow, additional SEMLS procedures may be needed to address new issues that arise, such as muscle tightness. Several studies have shown that these multilevel surgeries can improve walking ability. Saglam Y. et al., in 2016, studied the combination of femoral derotational osteotomy and soft tissue procedures in children with in-toeing gait. In 2022, Pierz K. et al. examined how SEMLS, including knee flexor lengthening combined with other techniques (such as triceps lengthening or tibial derotational osteotomy), improved walking in children with crouch gait. Moreira de Freitas Guardini K. et al., in 2021, also studied a large sample of children undergoing SEMLS, focusing on their clinical characteristics.

Evaluating the effects of surgery requires selecting appropriate outcome measures, which is not always simple. Most studies aim to improve "gait quality" but do not always confirm if the chosen parameters lead to real functional improvements for the patient. Some researchers use measures from physical exams (e.g., range of motion, muscle strength) or biomechanical data from gait analysis (3DGA, the gold standard for assessing gait in children with CP). These studies often focus on how the body moves (kinematics) and on spatiotemporal parameters such as walking speed and step length, along with summary indices. These parameters show changes in the specific area operated on and how the body moves as a whole. They provide information on alignment and symmetry of the legs during movement.

However, a well-aligned structure does not necessarily involve that the system works efficiently, meaning it minimizes energy expenditure during walking. Gait efficiency is especially important in children with CP, as many studies have shown that inefficient gait leads to increased energy consumption and mechanical work. Therefore, it is important to consider not only joint movement and overall performance but also other aspects, since kinematic data and physical exams do not provide information on gait efficiency.

Marconi V. et al. (2014) conducted a prospective study on energy consumption and mechanical work in children with CP after SEMLS. Their study showed a reduction in energy consumption after surgery, but the small sample size (10 children) and mixed group of patients (including hemiplegic, diplegic, and quadriplegic children) limit the generalizability of the results. Marconi V. et al. used the energy calculation method proposed by Willems P.A. et al. (1995), while Van de Walle P. et al. (2012) suggested that joint power calculations might be more valid and sensitive for CP. Other researchers have used indirect measures of efficiency, finding correlations between energy consumption and variables like pelvic vertical oscillation (assessed by the BEQ index, Kerrigan D.C. et al. 1996) or maximum knee and hip extension (Noorkoiv M. et al, 2019). These measures have been used to assess gait efficiency in CP, but not specifically to evaluate the effects of surgery.

The aim of this retrospective observational study is to describe the functional characteristics of children and adolescents with spastic cerebral palsy (CP) undergoing SEMLS and changes in their gait efficiency following surgery.

Methods:

This is a retrospective monocentric observational study. Outcome measures were collected before surgery (T0) and after surgery (T1) in a time span between 8 and 38 months. The surgical recommendation was tailored to the participants' requirements and decided through a comprehensive assessment, which included a standardized physical exam, radiographic studies, and instrumental gait analysis.

Gait analysis was performed by means of a Vicon® system (Oxford Metrics Group, Oxford, UK). The system was equipped with eight optoelectronic cameras, two force plates (AMTI, USA), and two video cameras. All assessments were conducted in the Motion Analysis Laboratory LAMBDA, Azienda USL-IRCCS di Reggio Emilia. The same assessor evaluated all participants.

Age and the level of Gross Motor Function Classification System (GMFCS) were collected before surgery.

The analyses will be conducted by the Statistics and Clinical Studies Office of the USL IRCCS in Reggio Emilia using SAS System, R, or SPSS software, depending on availability at the time. Quantitative and qualitative data will be analyzed and presented using mean, standard deviation (SD), median, interquartile range (IQR), and relative frequencies. Central tendency measures and percentages will be accompanied by 95% confidence intervals (CI). Normality of quantitative data will be assessed with the Shapiro-Wilk test. Appropriate statistical tests will be applied to compare measures between the two time points, T0 and T1.

To assess gait efficiency, the mean maximum extension values will be compared between T0 and T1 in the SEMLS surgery group using the paired Student's t-test or Wilcoxon test, depending on the normality assumption. Without aiming for comparison, the same measurements will also be described for the non-surgical group to observe trends.

For quantitative variable comparisons between the two time points, the paired Student's t-test or Wilcoxon test will be applied based on normality.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of diplegic or hemiplegic CP;
* GMFCS levels I, II, or III;
* aged between 4 and 20 years;
* Lower limb Single Event Multilevel Surgery (SEMLS)
* 3D gait analysis before and after surgery

Exclusion Criteria:

* more than one lower limb surgery event between the two gait assessments
* one single gait evaluation

Ages: 4 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will include patients who attended the Children Rehabilitation Unit of Local Health Authority of Reggio Emilia from 2011 to 2021. The study will focus on patients diagnosed with cerebral palsy who underwent lower limb SEMLS (single-event multilevel surgery) and 3D Gait Analysis before and after surgery.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
Mean maximum knee extension in the gait cycle | T0 (before SEML) and T1 (8-38 months after SEMLS)
  It is an indirect measure of walking efficiency. Greater knee extension leads to lower energy consumption.
  The measurement is calculated using 3D Gait Analysis. It has already been used to assess gait efficiency in children with CP (Noorkoiv, 2019), but never to evaluate the effects of surgery. These measures are useful when dynamic data are not available, such as when the stride length is short or the patient has low endurance, making it difficult to collect such data
change from baseline in maximum knee extension | T0 (before SEML) and T1 (8-38 months after SEMLS)
  It is an indirect measure of walking efficiency. Greater knee extension leads to lower energy consumption.
  The measurement is calculated using 3D Gait Analysis. It has already been used to assess gait efficiency in children with CP (Noorkoiv, 2019), but never to evaluate the effects of surgery. These measures are useful when dynamic data are not available, such as when the stride length is short or the patient has low endurance, making it difficult to collect such data.

SECONDARY OUTCOMES:
Correlation between the effect of surgery and the level of impairment | at T1( 8-38 months after SEMLS )
  Pearson's correlation will assess the relationship between age and surgical effect, measured as the difference in maximum knee extension. Additional correlation measures will be calculated to evaluate the relationship between surgical effect and the degree of impairment in patients.
Correlation between the effect of surgery and the age of participants | at T1( 8-38 months after SEMLS )
  Pearson's correlation will assess the relationship between age and surgical effect, measured as the difference in maximum knee extension. Additional correlation measures will be calculated to evaluate the relationship between surgical effect and the degree of impairment in patients
change from baseline in maximum hip extension | T0 (before SEML) and T1 (8-38 months after SEMLS)
  It is an indirect measure of walking efficiency. Greater knee extension leads to lower energy consumption.
  The measurement is calculated using 3D Gait Analysis. It has already been used to assess gait efficiency in children with CP (Noorkoiv, 2019), but never to evaluate the effects of surgery. These measures are useful when dynamic data are not available, such as when the stride length is short or the patient has low endurance, making it difficult to collect such data.
change from baseline in power produced by the ankle during push-off phase | at T1( 8-38 months after SEMLS )
  This parameter was chosen to assess efficiency because research shows that having adequate push-off strength is important for efficient walking (Jonkers et al., 2009). Keeping good propulsion ability after surgery is therefore a priority. Some authors have noted the risk of over-correction (Dietz et al., 2006; Sclavor et al., 2022), which can lead to iatrogenic weakness in the triceps and reduced walking efficiency (J. Lorentzen et al., 2020).
change from baseline in energy produced and absorbed | T0 (before SEML) and T1 (8-38 months after SEMLS)
  This parameter was chosen to assess efficiency because research shows that having adequate push-off strength is important for efficient walking (Jonkers et al., 2009). Keeping good propulsion ability after surgery is therefore a priority. Some authors have noted the risk of over-correction (Dietz et al., 2006; Sclavor et al., 2022), which can lead to iatrogenic weakness in the triceps and reduced walking efficiency (J. Lorentzen et al., 2020).
Change from baseline in Biomechanical Efficiency Quotient (BEQ) | T0 (before SEML) and T1 (8-38 months after SEMLS)
  To evaluate walking efficiency, the Biomechanical Efficiency Quotient (BEQ) (Kerrigan et al., 1996) was also included, obtained from three parameters: average step length, vertical displacement of the trunk during walking and height of the sacrum during standing. Kerrigan et al., show that this summary index is useful for evaluating the impact of physical therapy interventions, such as the use of Ankle Foot Orthosis (AFO), on biomechanical efficiency. From reviewing the literature, it appears that this measure has never been used to assess the effect of surgery.
Change from baseline in Gait Profile Score (GPS) | T0 (before SEML) and T1 (8-38 months after SEMLS)
  As a measure to evaluate gait quality, the Gait Profile Score (GPS) (Baker et al., 2009) was chosen. It is a general index that summarizes the overall deviation of kinematic gait data from reference data (Moreira de Freitas Guardini K. et al., 2021). The GPS can be broken down into the Gait Variable Score (GVS), which is based on nine kinematic variables: pelvic tilt, pelvic rotation, pelvic obliquity, hip and knee flexion/extension, ankle dorsiflexion/plantarflexion, hip abduction/adduction, hip rotation, and foot progression angle (Speciali DS et al., 2014).
  A decrease in the GPS score is considered an improvement. In the 2012 study, Baker et al. also defined the Minimal Clinical Important Difference (MCID), which is the smallest clinically relevant difference for this parameter. For the GPS, the MCID is 1.6°
Change from baseline in speed, Stride length, ratio frequency/stride lenght, stance time and double support | T0 (before SEML) and T1 (8-38 months after SEMLS)
  The spatiotemporal kinematic parameters will be used to compare overall walking performance, as done by other authors like Pierz et al. in 2022.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Sassi, MD, Principal Investigator — Azienda USL IRCCS of Reggio Emilia
Locations (2):
- Italy (2):
  - AziendaUSL IRCCS Reggio Emilia, Reggio Emilia
  - Azienda Unità Sanitaria Locale Reggio Emilia, Reggio Emilia

IPD SHARING:
Plan to Share IPD: No
To protect participant privacy the IPD will not be shared, unless upon reasonable request.

REFERENCES:
- [Background] Visscher R, Hasler N, Freslier M, Singh NB, Taylor WR, Brunner R, Rutz E. Long-term follow-up after multilevel surgery in cerebral palsy. Arch Orthop Trauma Surg. 2022 Sep;142(9):2131-2138. doi: 10.1007/s00402-021-03797-0. Epub 2021 Feb 23. PMID 33620528
- [Background] Vermuyten L, Desloovere K, Molenaers G, Van Campenhout A. Proximal femoral derotation osteotomy in children with CP : long term outcome and the role of age at time of surgery. Acta Orthop Belg. 2021 Mar;87(1):167-173. PMID 34129771
- [Background] Van de Walle P, Hallemans A, Schwartz M, Truijen S, Gosselink R, Desloovere K. Mechanical energy estimation during walking: validity and sensitivity in typical gait and in children with cerebral palsy. Gait Posture. 2012 Feb;35(2):231-7. doi: 10.1016/j.gaitpost.2011.09.012. Epub 2011 Oct 2. PMID 21962844
- [Background] van den Hecke A, Malghem C, Renders A, Detrembleur C, Palumbo S, Lejeune TM. Mechanical work, energetic cost, and gait efficiency in children with cerebral palsy. J Pediatr Orthop. 2007 Sep;27(6):643-7. doi: 10.1097/BPO.0b013e318093f4c3. PMID 17717464
- [Background] Schwartz MH, Rozumalski A, Novacheck TF. Femoral derotational osteotomy: surgical indications and outcomes in children with cerebral palsy. Gait Posture. 2014 Feb;39(2):778-83. doi: 10.1016/j.gaitpost.2013.10.016. Epub 2013 Oct 27. PMID 24268697
- [Background] Saglam Y, Ekin Akalan N, Temelli Y, Kuchimov S. Femoral derotation osteotomy with multi-level soft tissue procedures in children with cerebral palsy: Does it improve gait quality? J Child Orthop. 2016 Feb;10(1):41-8. doi: 10.1007/s11832-015-0706-4. Epub 2015 Nov 23. PMID 26597935
- [Background] Ries AJ, Schwartz MH. Low gait efficiency is the primary reason for the increased metabolic demand during gait in children with cerebral palsy. Hum Mov Sci. 2018 Feb;57:426-433. doi: 10.1016/j.humov.2017.10.004. Epub 2017 Oct 21. PMID 29066191
- [Background] Pierz K, Brimacombe M, Ounpuu S. Percutaneous hamstring lengthening in cerebral palsy: Technique and gait outcomes based on GMFCS level. Gait Posture. 2022 Jan;91:318-325. doi: 10.1016/j.gaitpost.2021.10.035. Epub 2021 Oct 29. PMID 34823200
- [Background] Palisano R, Rosenbaum P, Walter S, Russell D, Wood E, Galuppi B. Development and reliability of a system to classify gross motor function in children with cerebral palsy. Dev Med Child Neurol. 1997 Apr;39(4):214-23. doi: 10.1111/j.1469-8749.1997.tb07414.x. PMID 9183258
- [Background] Noorkoiv M, Lavelle G, Theis N, Korff T, Kilbride C, Baltzopoulos V, Shortland A, Levin W, Ryan JM. Predictors of Walking Efficiency in Children With Cerebral Palsy: Lower-Body Joint Angles, Moments, and Power. Phys Ther. 2019 Jun 1;99(6):711-720. doi: 10.1093/ptj/pzz041. PMID 31155663
- [Background] de Freitas Guardini KM, Kawamura CM, Lopes JAF, Fujino MH, Blumetti FC, de Morais Filho MC. Factors related to better outcomes after single-event multilevel surgery (SEMLS) in patients with cerebral palsy. Gait Posture. 2021 May;86:260-265. doi: 10.1016/j.gaitpost.2021.03.032. Epub 2021 Mar 27. PMID 33813186
- [Background] Moisan G, Bonnefoy-Mazure A, De Coulon G, Tabard-Fougere A, Armand S, Turcot K. Assessment of gait quality and efficiency after undergoing a single-event multilevel surgery in children with cerebral palsy presenting an intoeing gait pattern. Childs Nerv Syst. 2022 Aug;38(8):1523-1530. doi: 10.1007/s00381-022-05548-x. Epub 2022 May 12. PMID 35552497
- [Background] Marconi V, Hachez H, Renders A, Docquier PL, Detrembleur C. Mechanical work and energy consumption in children with cerebral palsy after single-event multilevel surgery. Gait Posture. 2014 Sep;40(4):633-9. doi: 10.1016/j.gaitpost.2014.07.014. Epub 2014 Jul 24. PMID 25107323
- [Background] Kruger KM, Constantino CS, Graf A, Flanagan A, Smith PA, Krzak JJ. What are the long-term outcomes of lateral column lengthening for pes planovalgus in cerebral palsy? J Clin Orthop Trauma. 2021 Nov 26;24:101717. doi: 10.1016/j.jcot.2021.101717. eCollection 2022 Jan. PMID 34926149
- [Background] Kerrigan DC, Thirunarayan MA, Sheffler LR, Ribaudo TA, Corcoran PJ. A tool to assess biomechanical gait efficiency; a preliminary clinical study. Am J Phys Med Rehabil. 1996 Jan-Feb;75(1):3-8. doi: 10.1097/00002060-199601000-00003. PMID 8645436
- [Background] Kadhim M, Miller F. Crouch gait changes after planovalgus foot deformity correction in ambulatory children with cerebral palsy. Gait Posture. 2014 Feb;39(2):793-8. doi: 10.1016/j.gaitpost.2013.10.020. Epub 2013 Nov 2. PMID 24316233
- [Background] Almoajil H, Dawes H, Hopewell S, Toye F, Jenkinson C, Theologis T. Development of a core outcome set for lower limb orthopaedic surgical interventions in ambulant children and young people with cerebral palsy: a study protocol. BMJ Open. 2020 Mar 4;10(3):e034744. doi: 10.1136/bmjopen-2019-034744. PMID 32139490
- [Background] Graham HK, Rosenbaum P, Paneth N, Dan B, Lin JP, Damiano DL, Becher JG, Gaebler-Spira D, Colver A, Reddihough DS, Crompton KE, Lieber RL. Cerebral palsy. Nat Rev Dis Primers. 2016 Jan 7;2:15082. doi: 10.1038/nrdp.2015.82. PMID 27188686
- [Background] Dohin B, Haddad E, Zagorda-Pallandre B, Zemour M. Outcomes of isolated soft tissue surgery for in-toeing gait in patients with ambulatory cerebral palsy. Orthop Traumatol Surg Res. 2020 Nov;106(7):1367-1371. doi: 10.1016/j.otsr.2020.06.008. Epub 2020 Sep 29. PMID 33008781